CLINICAL TRIAL: NCT01255566
Title: A Comparison of Medical Therapy to Medical Therapy Plus Endoscopic Sinus Surgery in Patients With Chronic Rhinosinusitis
Brief Title: Medical Therapy Versus Sinus Surgery for Chronic Rhinosinusitis: A Prospective, Multi-institutional Study
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Medical University of South Carolina (Other); Northwestern University (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Dr. Timothy L. Smith, Professor, Oregon Health and Science University
Other Study IDs: unfunded
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Rhinosinusitis; Sinusitis
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Medical therapy cohort: For patients electing continued medical therapy, medication was prescribed based on the disease process and the judgment of the treating rhinologist. Treatment was not specifically dictated or prescribed by the study protocol.
- Surgical cohort: For patients electing ESS, surgery was performed by the enrolling rhinologist. In addition, medical management was administered in the perioperative and postoperative periods as dictated by the disease process and the judgment of the treating rhinologist. Treatment was not specifically dictated or prescribed by the study protocol.

SUMMARY:
This investigation is a prospective, multi-institutional cohort study comparing the differences in health-related quality-of-life (HRQoL) improvements between subjects electing continued medical management for chronic rhinosinusitis and those electing medical management plus surgical intervention.

Our hypothesis is 3 fold: 1. That patients electing continued medical management will have less disease severity as measured by CT and baseline HRQoL scores, 2. Patients undergoing medical management plus ESS for chronic rhinosinusitis will experience a larger improvement in health related quality of life (HRQoL)compared to patients electing medical management alone, and 3. Patients undergoing medical management plus ESS for chronic rhinosinusitis will use fewer antibiotics, systemic steroids, and miss fewer days of work/school compared to patients electing medical management alone.

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS) is a common health condition in the United States resulting in more than 500,000 surgical procedures annually. Since CRS is a disease process that is known to adversely affect quality of life, it is important to understand the short-term and long-term implications of different treatment options as documented by our patients' perception of their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>= 18 years old)
* Diagnosed with chronic rhinosinusitis
* Failed medical management to date
* Self-selected either sinus surgery or continued medical therapy as next treatment option
* Able to complete surveys in English

Exclusion Criteria:

* Unable to complete surveys in English
* Children (< 18 years old)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects (> 18 years) were prospectively enrolled from four tertiary rhinology practices including Oregon Health & Science University (OHSU); Northwestern University (NWU); Medical University of South Carolina (MUSC); and the University of Pennsylvania (UPenn). All patients were diagnosed with chronic rhinosinusitis (CRS) as defined by the 2007 Adult Sinusitis Guidelines.
Sampling Method: Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2009-08; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Rhinosinusitis Disability Index and Chronic Sinusitis Survey | Change from baseline to 12 months
  The RSDI is a validated, disease-specific quality-of-life survey designed for patients with sinonasal disease. The RSDI has three separate subscales incorporating 30 questions with a total score range of 0-120. The CSS is a validated, 6 question survey with two separate subscales which measure the impact of sinonasal symptoms and medication use in the preceding 8-week period. Total score range of 0-100 for total and subscale measures.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- [Derived] Smith TL, Kern R, Palmer JN, Schlosser R, Chandra RK, Chiu AG, Conley D, Mace JC, Fu RF, Stankiewicz J. Medical therapy vs surgery for chronic rhinosinusitis: a prospective, multi-institutional study with 1-year follow-up. Int Forum Allergy Rhinol. 2013 Jan;3(1):4-9. doi: 10.1002/alr.21065. Epub 2012 Jun 26. PMID 22736422
- [Derived] Smith TL, Kern RC, Palmer JN, Schlosser RJ, Chandra RK, Chiu AG, Conley D, Mace JC, Fu RF, Stankiewicz JA. Medical therapy vs surgery for chronic rhinosinusitis: a prospective, multi-institutional study. Int Forum Allergy Rhinol. 2011 Jul-Aug;1(4):235-41. doi: 10.1002/alr.20063. Epub 2011 Jun 6. PMID 22287426